CLINICAL TRIAL: NCT04521972
Title: Impact of Light on Labor Progression
Brief Title: Impact of Room Light on Uterine Contractions and Labor Progression in Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: McLaren Health Care (Other)
Responsible Party: Principal Investigator, Hanne M Hoffmann, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00003410
Record Dates: First submitted 2020-08-13; First posted 2020-08-21 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy Related; Labor; Poor; Uterine Contractions Weak

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Group 1 (Active Comparator): Natural non-augmented labor with room lights ON. This is what is currently done in the hospital, and thus does not change any current medical practices.
  Interventions: Device: Room light/light bulb
- Group 2 (Active Comparator): Augmented labor with room lights ON. This group will be a subgroup of Group 1 (Natural non-augmented labor with room lights ON), as labor-augmentation cannot be planned for until the patient is in labor or labor needs to be augmented for medical reasons.
  Interventions: Device: Room light/light bulb
- Group 3 (Experimental): Natural non-augmented labor with reduced or red room lights.
  Interventions: Device: Room light/light bulb
- Group 4 (Experimental): Augmented labor with reduced or red room lights. This group will be a subgroup of Group 3, as augmented labor cannot be planned for until the patient is in labor or labor needs to be augmented for medical reasons.
  Interventions: Device: Room light/light bulb

INTERVENTIONS:
Device: Room light/light bulb — Room light will be ON/OFF or red light used in the room. Reducing/eliminating light in the room in the evening and night is expected to allow the natural release of melatonin, which is thought to promote uterine contractions in late pregnancy.

SUMMARY:
Today it remains a challenge to successfully both halt and induce labor progression. Induction of labor is a common obstetric intervention that 1 in 4 women will experience. The goal of induction of labor is to achieve a vaginal birth, however in almost 40% of first-time mothers it fails. Failed labor inductions require a caesarean delivery, which is associated with a vast range of adverse effects for both the mother and her baby. In this application we propose that a simple manipulation of room light will increase the success of vaginal birth through the use of optimal room light settings (halting labor=lights ON, promoting labor=reduced room light/red room light).

A sparse literature has shown that the hormone melatonin might be an important hormone to consider during late pregnancy and labor. Pineal melatonin release is only released in darkness at night, where nocturnal light such as room light, suppress pineal melatonin release, reducing uterine contractions (Olcese et al 2013, https://pubmed.ncbi.nlm.nih.gov/22556015/, Rahman et al 2019, https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6453747/). Melatonin receptor become upregulated in the pregnant myometrium (uterine smooth muscle), and a small study in women having preterm birth, showed a high expression of melatonin receptor, at a gestational week where women not having preterm uterine contractions, had low levels of melatonin receptor, suggesting that premature increase in myometrium melatonin receptor might in some women be associated with preterm labor and birth (Olcese et al 2013, https://pubmed.ncbi.nlm.nih.gov/22556015/).

This study will address how room light impacts melatonin release and uterine contractions in healthy pregnant women.

DETAILED DESCRIPTION:
Overview of study layout

The indicated prenatal visit weeks are approximate time points. The prenatal visit only needs to occur prior to the sample collection time point.

Time point 1 (First interaction with patient). First trimester of pregnancy. Recruiting patients who have an Ob/Gyn appointment to start prenatal care. During this visit we will recruit women with confirmed pregnancy into the study. During the meeting with the Ob/Gyn, the study goals and layout of study will be explained to the patient. The patient will not be informed about the expected outcome of nocturnal light on uterine contractions and labor progression.

The patient will be provided with the consent forms and given time to read and ask questions about the forms prior to signing. If the patient desires to read the consent form at home, and enroll later, that is also possible.

After enrolling in the study, the patient will be given the below information to complete during week 11 of pregnancy in their home:

1. Sleep, activity and saliva sample questionnaires (printout).
2. Tubes and cooler to collect two saliva samples at home:

   1. Sample 1 is collected 0-3h after sunset
   2. Sample 2 is collected 0-3h after sunset in darkness
   3. Sample 3 is collected 0-3h after sunset with lights ON
3. Note: Questionnaires are filled on the day of saliva collection. Patients will return the frozen saliva samples and questionnaires at their next in person Ob/Gyn visit or when they come to the Hoffmann laboratory in the third trimester.

Time point 2. Week 20-22 of pregnancy, in person Ob/Gyn prenatal care visit.

During visit with Ob/Gyn the patient will be given the below information to complete during week 20-22 of pregnancy in their home:

1. Sleep, activity and saliva sample questionnaires (printout).
2. Tubes and cooler to collect two saliva samples at home:

   1. Sample 1 is collected 0-3h after sunset
   2. Sample 2 is collected 0-3h after sunset in darkness
   3. Sample 3 is collected 0-3h after sunset with lights ON
3. Note: Questionnaires are filled in the day of saliva collection. Patients will return the frozen saliva samples and questionnaires at their next in person Ob/Gyn visit or when they come to the Hoffmann laboratory in the third trimester.

Time point 3. Week 28 of pregnancy-assigning patients into study groups. During the prenatal visit around week 28, the desired birth plan will be discussed with the patient. During this meeting, the patient will not know what group they are assigned, nor how we expect the light conditions to impact labor progression. The primary goal of this discussion is to determine if the patient is anticipating a planned C-section.

The five study groups patients are assigned to are as follows:

Group 1: Natural non-augmented labor with room lights ON. This is what is currently done in the hospital, and thus does not change any current medical practices.

Group 2: Augmented labor with room lights ON. This group will be a subgroup of Group 1, as labor-augmentation cannot be planned for until the patient is in labor or labor needs to be augmented for medical reasons.

Group 3: Natural non-augmented labor with reduced or red room lights. Group 4: Augmented labor with reduced or red room lights. This group will be a subgroup of Group 3, as augmented labor cannot be planned for until the patient is in labor or labor needs to be augmented for medical reasons.

Group 5: C-section. Scheduled and emergency C-sections. Uterine samples will be collected in this group for ex vivo studies.

Group assignments will be achieved through randomization as follows.

1. Women anticipating a C-section are assigned to group 5.
2. Women anticipating a vaginal birth are randomly assigned to Group 1 and Group 3. This will allow to have ½ women going through labor with lights ON, and ½ the women going through labor with reduced room lights.

Note On a monthly basis, we will evaluate the number of women who have given birth in Groups 1-5. Based on this we will readjust group assignments of women entering the study, to assure comparable group sizes in groups 1-5 to the greatest degree possible.

Time point 4. Third trimester: Weeks 32-34 of pregnancy We will schedule 2 appointments during weeks 32-34 of pregnancy where the women are able to come to the Hoffmann laboratory at MSU. One appointment will take place around sunset and be of a duration of 2-3h, starting around 7-8PM. The second appointment will take place in the morning between 8AM and 12PM. This appointment will be of ~ 90 min.

During each of these visits at the Hoffmann laboratory the study participants will:

1. Be placed in the study room with a specific room light condition (bright white light or dim red light).
2. Study participants will fill out the sleep, activity and saliva sample questionnaires.
3. Study participants will have their uterine contractions measured for 60 min at the morning appointment and for 120-150 min at the evening appointment.

For details of this visit see Annex 1 (last page of this document)

Time point 5. Third trimester: Weeks 38-40 We will schedule 2 appointments during weeks 38-40 of pregnancy where the women are able to come to the Hoffmann laboratory at MSU. One appointment will take place around sunset and be of a duration of 2-3h, starting around 7-8PM. The second appointment will take place in the morning between 8AM and 12PM. This appointment will be of ~ 90 min.

During each of these visits at the Hoffmann laboratory the study participants will:

1. Be placed in the study room with a specific room light condition (bright white light or dim red light).
2. Study participants will fill out the sleep, activity and saliva sample questionnaires.
3. Study participants will have their uterine contractions measured for 60 min at the morning appointment and for 120-150 min at the evening appointment.

For details of this visit see Annex 1 (last page of this document)

Time point 6. Evaluate labor progression and duration in rooms with lights ON and reduced light.

When the study participant is admitted to the hospital in labor, the following steps will be done:

* Room light will be adapted as indicated in patient chart, and room light-intensity measured.
* Continuously record uterine contractions.
* Collect saliva sample at admission, and every 2 h thereafter until 6h after birth.

Additional steps for women having a C-section When a woman is scheduled to have a C-section (planned or emergency), Dr. Hoffmann is notified by phone or text to 858 344 8389 at the time of C-section scheduling. After delivery of the infant by C-section and removal of the placenta, a full-thickness myometrial sample is removed from the superior edge of the transverse uterine incision. The wedge-shaped sample, obtained by sharp dissection with a curved Mayo scissors, is approximately 1 cm wide and 5 cm long. The samples will immediately be placed in sterile containers and collected by a Hoffmann laboratory member for transport to MSU where they will be stored in the -80C freezer and used for uterine contraction analysis The myometrium sample is placed in a deidentified numbered tube and handed over to experimenter to allow processing. Dr. Hoffmann or a participating Hoffmann laboratory member will come to the hospital to collect the myometrium sample within 90 min after C-section completion.

In home delivery In the scenario of home delivery, all data points prior to delivery will be included in the study. Home delivery will only impact the last study time point, as all data collections prior to delivery are the same for all the study groups.

ELIGIBILITY:
Inclusion criteria:

* Are pregnant
* Are 18-42 years old
* Medically cleared for participation by Medical Investigator
* Willingness to allow the study access to information in the participant's medical record
* Willingness to be notified of incidental findings from study procedures
* Willingness to measure and report on lighting conditions during specified time periods
* Willingness to use a uterine contraction home monitor system, and report results
* Willingness to adapt lighting during studies in home and/or hospital
* Willingness to wear blue-filter glasses if requested
* Willingness to report use of melatonin (for sleep)
* Willingness to stop melatonin use if requested

Exclusion criteria

* Pre-pregnancy BMI >36kg/m2
* HIV or AIDS (self-reported)
* Severe anemia (hemoglobin <8g/dL and/or hematocrit <24%)
* History or current psychotic disorder or diagnosis of a current major depressive episode or bipolar disorder
* Current use of one or more of the following medications: metformin, systemic steroids, antipsychotic agents (e.g., Abilify, Haldol, Risperdal, Seroquel, Zyprexa), anti-seizure medications or mood stabilizers that would be expected to have a significant impact on body weight (e.g., Depakote, Lamictal, Lithium, Neurontin, Tegretol, Topamax, Keppra), medications for ADHD including amphetamines and methylphenidate
* Continued use of weight loss medication including OTC and dietary supplements for weight loss (e.g., Adipex, Suprenza, Tenuate, Xenical, Alli, conjugated linoleic acid, Hoodia, Green tea extract, Guar gum, HydroxyCut, Sensa, Corti-slim, Chromium, chitosan, Bitter orange) Other Exclusion Criteria
* Recent history of or currently smoking, drinking alcohol or abusing drugs (prescription or recreational)
* Plans to move out of the study area within the next year or plans to be out of the study area for more than 8 weeks in the next 12 months
* Planned termination of pregnancy

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study is focused on pregnancy and labor, as such only women are include in the study.
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Nocturnal room light changes uterine contractions in pregnant women | From confirmation of pregnancy till birth. The study time frame is up to 40 weeks.
  We will measure how room light during day and night periods impact uterine contractions during pregnancy and labor.

SECONDARY OUTCOMES:
Nocturnal room light changes melatonin release in pregnant women | From confirmation of pregnancy till birth. The study time frame is up to 40 weeks.
  We will measure how room light during day and night periods change melatonin release during pregnancy and labor.

CONTACTS AND LOCATIONS:
Overall Officials: Hanne M Hoffmann, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
  Identified and de-identified data will not be used or shared for commercial profit.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.